CLINICAL TRIAL: NCT00497120
Title: A Combined Surgical and Medical Approach in Mild Sleep Apnea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC 2/27/99
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; snoring; acetazolamide; uvulopalatopharyngoplasty; daytime sleepiness; upper airway
MeSH Terms: conditions — Sleep Apnea Syndromes; Snoring; Disorders of Excessive Somnolence | interventions — Acetazolamide

INTERVENTIONS:
Drug: acetazolamide
Drug: placebo
Procedure: uvulopalatopharygoplasty

SUMMARY:
The aim of the study is to investigate wether the adjuvant (postoperative) administration of acetazolamide can improve the surgical results after uvulopalatopharyngoplasty in patients with mild sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* 5 ≤ Apnea Hypopnea Index (AHI) < 20
* Socially disturbing snoring: Visual Analogue Scale (VAS)snoring > 6/10
* Based on clinical examination and polysomnography, patient is regarded eligible for uvulopalatopharyngoplasty (UPPP)

Exclusion Criteria:

* Previous surgical treatment for sleep-disordered breathing.
* Periodic Limb Movement Disorder (PLMD) with arousals and other reasons possibly explaining the Excessive Daytime Sleepiness (EDS) based on Epworth Sleepiness Scale (ESS).
* Forced expiratory volume in 1 second (FEV1) < 80 % pred.
* Echocardiography: ejectionfraction < 35 % or dyastolic dysfunction grade 2 or more.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Polysomnographic parameters

SECONDARY OUTCOMES:
subjective sleepiness
subjective snoring
satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium